CLINICAL TRIAL: NCT03109223
Title: Effects of Addition to Infant Formula of 2-fucosyllactose (2-FL) on Growth, Fecal Bacterial Populations and Safety
Brief Title: Addition to Infant Formula of 2-fucosyllactose (2-FL)
Acronym: 2-FL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PBM Nutritionals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PRG-VA-17-001
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Growth of Infants

STUDY DESIGN:
Intervention Model Description: Double-blind randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Commercially availabel infant formula (Active Comparator)
  Interventions: Other: sole source nutrition
- Test formula with 2-FL (Experimental)
  Interventions: Other: sole source nutrition
- Breast Fed (Active Comparator)
  Interventions: Other: sole source nutrition

INTERVENTIONS:
Other: sole source nutrition — Infant formula

SUMMARY:
OBJECTIVES:

Primary:

The primary objective is to determine whether the mean weight gain over a 16-week interval starting on or before 14 days of life differs between infants fed one of two infant formulas as their sole source of nutrition: a commercial formula using a canola l fat blend (Control, E23) or the same formula containing the human milk oligosaccharide (Test (HMO) 2-fucosyllactose (2FL). Mean weight gain also will be compared to that of a concurrently enrolled reference group of exclusively breastfed infants.

DETAILED DESCRIPTION:
METHODOLOGY/ STUDY DESIGN: This study is double blinded-randomized controlled trial with two arms and a reference breast fed group. The experimental variable is the composition of infant formula fed to healthy term infants for a period of 16 weeks upon entering the study as their sole source of nutrition. The formulations are a commercial control (Control, NPS-E23); and the control formula containing the human milk oligosaccharide (HMO) 2-fucosyllactose (2FL) at 1g/L (HMO, NPS-E23XA).

Infants will be enrolled on or before 14 days of age and fed a study assigned formula for 16 weeks. Weight, length and head circumference will be measured at baseline and 2, 4, 6, 8, 12 and 16 weeks of study entry. Formula volume will be recorded for a three-day period before each visit. Fecal samples will be obtained at baseline (convenience samples) and at week 16 for all subjects and analyzed for microbial populations. Buccal cheek cells of all infants, and mothers of breast fed infants, obtained by swab at week 16 will be genotyped for FUT2. Information on adverse events and new/change of medications will be collected at in person visits and by telephone interviews between in-person visits.

NUMBER OF SUBJECTS: It is estimated that approximately up to approximately 200 subjects will be enrolled in the formula groups to obtain up to approximately 65 evaluable per protocol subjects in each group. As non-randomized reference group of approximately 85 breastfed infants will be enrolled to obtain approximately 65 evaluable infants.

ELIGIBILITY:
Inclusion Criteria:

* 1. At birth:

  * Healthy, term (37-42 weeks), appropriate for gestational age 2. At the time of enrollment:
  * < 14 days post-natal age at time of enrollment, either gender
  * Exclusively formula fed or breastfed upon enrollment Subject must be in general good health and free from any clinically significant disease, condition, or illness that might interfere with the study evaluations. Prior labs must be present to confirm good health.
  * Formula group infants: Mother has determined to use infant formula exclusively for feeding her baby through at least 16 weeks.
  * Reference breastfed infants: Mother has determined to breastfeed exclusively through at least 16 weeks Written informed consent of parent/guardian, prior to any study related procedures being performed.

Exclusion Criteria:

* 1. Any clinically significant abnormal findings, as determined by the investigator, on the subject's medical history or physical exam during screening.

  2. Use of systemic medications by the subject that in the Investigator's opinion could impact evaluation of the subject's assessments.

  3. Discontinuation of exclusive breastfeeding by reference group (breastfed) infants.

  4. Fed with baby/solid foods on average more than once per day.

Ages: 4 Days to 36 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 221 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Growth | 4 months
  Growth as compared to WHO Growth Charts

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Qualmedica Research, LLC dba Pedia Research, LLC, Evansville, Indiana
  - Advantage Clinical Trials, The Bronx, New York
  - JBR Clinical Research, Salt Lake City, Utah
  - PI-Coor Clinical Research, LLC, Burke, Virginia
- Hospital Clinica Bendana, San Pedro Sula, Honduras

IPD SHARING:
Plan to Share IPD: Undecided